CLINICAL TRIAL: NCT01041573
Title: Safety and Immunogenicity of the Japanese Encephalitis Vaccine IC51 (IXIARO®) in a Pediatric Population. Open Label, Randomized, Active Controlled, Phase 3 Study
Brief Title: Safety and Immunogenicity of the Japanese Encephalitis Vaccine IC51 (IXIARO®) in a Pediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IC51-323
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Encephalitis
Keywords: Pediatric; Japanese Encephalitis Vaccine; endemic countries; to assess the systemic and local safety profile of purified inactivated Japanese Encephalitis Virus (JEV) vaccine IC51
MeSH Terms: conditions — Encephalitis | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IC51 0.5 mL (Experimental): Japanese Encephalitis Vaccine 6mcg im. at day 0 and day 28
  Interventions: Biological: IC51 Japanese Encephalitis
- IC51 0.25 mL (Experimental): Japanese Encephalitis Vaccine 3mcg im. at day 0 and day 28
  Interventions: Biological: IC51 Japanese Encephalitis
- Havrix 720 (Active Comparator): Havrix®720 0.5 ml im. at day 0 and month 7
  Interventions: Biological: Havrix®720
- Prevnar (Active Comparator): Prevnar 0.5 ml im. at day 0 and day 56 and month 7 or 0.5 ml im. at day 0, day 28 and day56 and month 7-13
  Interventions: Biological: Prevnar

INTERVENTIONS:
Biological: IC51 Japanese Encephalitis — 6 mcg or 3 mcg im. at day 0 and day 28
  Arms: IC51 0.25 mL; IC51 0.5 mL
Biological: Havrix®720 — 0.5 ml im. at day 0 and month 7
  Arms: Havrix 720
Biological: Prevnar — 0.5 ml im. at day 0 and day 56 and month 7
  Arms: Prevnar

SUMMARY:
The primary objective is to assess the systemic and local safety profile of purified inactivated Japanese Encephalitis Virus (JEV) vaccine IC51 administered in two doses in a 28 days interval up to Month 7 after the first IC51 vaccination in a pediatric population from endemic regions.

DETAILED DESCRIPTION:
Open-label, randomized, active controlled Phase 3 study in children aged ≥ 2 months to < 18 years. Subjects aged ≥ 2 months to < 12 months were randomized in a 2:1 ratio to receive IC51 (0.25 ml dose) or Prevnar® as a safety comparator. Children aged ≥ 12 months to < 3 years and ≥ 12 years to < 18 years were randomized in a 3:1 ratio to receive IC51 (0.25 ml dose < 3 years, 0.5 ml ≥ 12 years) or HAVRIX®720 as safety comparator.

For subjects aged ≥ 3 years to < 12 years, a dose finding run-in phase was performed. A total of 200 subjects were randomized 1:1 to receive either the 0.25 ml or the 0.5 ml dose of IC51, and the appropriate dose was determined based on an interim analysis. After this run-in phase, 300 further children in this age group were randomized 2:1 to receive either 0.5 ml of IC51 or HAVRIX®720.

Immunogenicity was be studied in a subgroup of 30 children aged ≥ 2 months to < 12 months; 125 children aged ≥ 12 months to < 3 years and 140 children ≥ 12 years to < 18 years. For the age group of ≥ 3 to < 12 years immunogenicity was assessed in the 200 children enrolled during the dose-finding run-in phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy children and adolescents aged > 2 months to < 18 years at the time of first vaccination.
* Written informed consent by the subject's legal representative(s), according to local requirements, and written informed assent of the subject, if applicable.
* Female subjects: either no childbearing potential or negative pregnancy test, for females after menarche willingness to practice a reliable method of contraception.

Exclusion Criteria:

* Clinical manifestation of Japanese Encephalitis
* History of Flavivirus vaccination (including any investigational vaccines)
* History of vaccination with HAVRIX®720 and/or Prevnar®
* History of immunodeficiency or immunosuppressive therapy
* Known HIV, HBV or HCV infection
* History of hypersensitivity reactions to other vaccines
* Acute febrile infection at each visit during which the subject receives a vaccination
* Active or passive immunization within 2 weeks prior to the first IC51 vaccination and up to the second IC51 vaccination.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1869 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Kadlecek, Study Director — Valneva Austria GmbH
Locations (2):
- Philippines (2):
  - Research Institute for Tropical Medicine, City of Muntinlupa, Filinvest Corporate City
  - Department of Pediatrics, UP-Philippine General Hospital, Manila

RESULTS

PARTICIPANT FLOW:
Groups:
- IC51 0.5 mL: Japanese Encephalitis Vaccine 6mcg i.m. at day 0 and day 28
- IC51 0.25 mL: Japanese Encephalitis Vaccine 3mcg i.m. at day 0 and day 28
- Havrix 720: Havrix®720 0.5 ml i.m. at day 0 and month 7
- Prevnar: Prevnar 0.5 ml i.m. at day 0 and day 56 and month 7 or 0.5 ml i.m. at day 0, day 28 and day 56 and month 7-13
Period: Overall Study
Arm/Group | IC51 0.5 mL | IC51 0.25 mL | Havrix 720 | Prevnar
Started | 540 | 871 | 394 | 64
Completed | 535 | 858 | 387 | 62
Not Completed | 5 | 13 | 7 | 2
Not completed — Withdrawal by Subject | 2 | 5 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — relocation | 1 | 4 | 3 | 1
Not completed — further blood extraction | 0 | 1 | 0 | 0
Not completed — positive to anti-HCV | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prevnar: Prevnar 0.5 ml i.m. at day 0 and day 56 and month 7 or 0.5 ml i.m. at day 0, day 28 and day56 and month 7-13
- Total: Total of all reporting groups
Arm/Group | IC51 0.25 mL | IC51 0.5 mL | Havrix 720 | Prevnar | Total
Number analyzed (Participants) | 871 | 540 | 394 | 64 | 1869
Age, Customized [Number; unit: participants]
  2 months - < 1 year | 131 | 0 | 0 | 64 | 195
  1 year - < 3 years | 640 | 0 | 213 | 0 | 853
  3 years - < 12 years | 100 | 300 | 101 | 0 | 501
  12 years - < 18 years | 0 | 240 | 80 | 0 | 320
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 449 | 249 | 197 | 30 | 925
  Male | 422 | 291 | 197 | 34 | 944
Region of Enrollment [Number; unit: participants]
  Philippines | 871 | 540 | 394 | 64 | 1869

OUTCOME MEASURES:

1. Primary Outcome: Rate of Subjects With Serious Adverse Events and Medically Attended Adverse Events Until Day 56 After First Vaccination
Description: Rate of subjects with these types of AEs, comparison vs respective control vaccine stratified by age group: All study participants aged < 1 year: IC51 0.25mL vs. Prevnar; All study participants aged 1 year and above: IC51 0.25 mL or =.5 mL vs. Havrix.
Time Frame: until Day 56
Population: As specified per protocol, safety parameters were compared between treatment groups (i.e. IC51 any dose level versus Havrix or Prevnar), stratified by age. Age was the determining factor of the respective safety comparators Prevnar (<1yrs) and HAVRIX (1+ yrs). Different dose levels of IC51 were grouped for these analyses, to test the hypothesis that events do not occur in higher frequency after vaccination with IC51 compared to vaccination with Prevnar® or Havrix®720.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- IC51, Subjects Aged >= 1 Year: IC51 Japanese Encephalitis: 6 mcg or 3 mcg im. at day 0 and day 28
- Havrix 720: Havrix®720 0.5 ml im. at day 0 and month 7; active comparator for subjects aged > 1 year
- IC51, Subjects Aged >= 2 Months to <1 Year: Japanese Encephalitis Vaccine 3mcg im. at day 0 and day 28
- Prevnar: Active comparator in subjects aged ≥ 2 months to < 1 year:
  * Subjects aged ≥ 2 to < 6 months: 4 intramuscular vaccinations, Days 0, 28, 56 and Month 7-13 (subjects aged ≥ 2 to < 6 months were to receive the fourth Prevnar® vaccination when 12-15 months old, i.e., the vaccination was to be performed outside the study, depending on the subject´s age at day of first vaccination).
  * Subjects aged ≥ 6 months to < 1 year: 3 intramuscular vaccinations, Days 0, 56 and Month 7.
Arm/Group | IC51, Subjects Aged >= 1 Year | Havrix 720 | IC51, Subjects Aged >= 2 Months to <1 Year | Prevnar
Number analyzed (Participants) | 1280 | 394 | 131 | 64
percentage of participants | 16.1 [14.1 to 18.2] | 14.2 [10.9 to 18.1] | 38.2 [29.8 to 47.1] | 42.2 [29.9 to 55.2]
Statistical Analysis 1: Comparison: IC51, Subjects Aged >= 2 Months to <1 Year vs Prevnar; Test type: Superiority or Other; p = 0.641, Fisher Exact
Statistical Analysis 2: Comparison: IC51, Subjects Aged >= 1 Year vs Havrix 720; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Geometric Mean Titers (GMT) for JEV Neutralizing Antibodies
Description: GMT for JEV neutralizing antibodies is presented per dose group rather than age group due to overlapping age groups. IC51 0.25 mL includes subjects aged 2 months to < 12 years; IC51 0.5 mL includes subjects aged ≥ 3 years to < 18 years.
Time Frame: Day 0, 56 and at Month 7
Population: Intent-to-treat Population: all subjects randomized into the immunogenicity subgroup, who received at least 1 vaccination. Subjects were analyzed according to the treatment group to which they were randomized rather than by the actual vaccine they received.
Measure: Geometric Mean (Standard Deviation); unit: Geometric Mean Titer
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 255 | 241
Geometric Mean Titer
  Day 0 | 5.79 (1.802) | 9.78 (2.944)
  Day 56 | 199.39 (3.387) | 190.77 (2.747)
  Month 7 | 37.99 (3.267) | 64.83 (3.242)

3. Secondary Outcome: Seroconversion Rate (SCR) at Days 0, 56 and at Month 7
Description: Seroconversion was defined as a PRNT50 titer of at least 1:10. SCRs are presented per dose group rather than age group due to overlapping age groups. IC51 0.25 mL includes subjects aged 2 months to < 12 years; IC51 0.5 mL includes subjects aged ≥ 3 years to < 18 years.
Time Frame: Days 0, 56 and at Month 7
Population: "number analyzed" is dependent on number of serum samples available for testing
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 255 | 241
percentage of participants
  Day 0: number analyzed (Participants) | 254 | 241
  Day 0 | 7.5 [4.8 to 11.4] | 33.6 [27.9 to 39.8]
  Day 56: number analyzed (Participants) | 246 | 237
  Day 56 | 98.0 [95.3 to 99.1] | 100.0 [98.4 to 100.0]
  Month 7: number analyzed (Participants) | 248 | 237
  Month 7 | 83.9 [78.8 to 87.9] | 94.5 [90.8 to 96.8]

4. Secondary Outcome: Rate of Subjects With SAEs and Medically Attended AEs
Description: Rate of subjects with SAEs and medically attended AEs; For this analysis IC51 vaccine recipients are displayed by age group rather than by dose group. This allows comparison of the safety profile of IC51 with the active control for the respective age group: Prevnar for study participants aged >= 2 months to <1 year and Havrix 720 for study participants aged >= 1 year.
Time Frame: up to Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Havrix 720: Havrix®720 0.5 ml im. at day 0 and month 7; active comparator for subjects aged ≥1 to <18 years
- Prevnar: Active comparator for subjects < 1 year of age:
  * Subjects aged ≥ 2 to < 6 months: 4 intramuscular vaccinations, Days 0, 28, 56 and Month 7-13 (subjects aged ≥ 2 to < 6 months were to receive the fourth Prevnar® vaccination when 12-15 months old, i.e., the vaccination was to be performed outside the study, depending on the subject´s age at day of first vaccination).
  * Subjects aged ≥ 6 months to < 1 year: 3 intramuscular vaccinations, Days 0, 56 and Month 7.
Arm/Group | IC51, Subjects Aged >= 1 Year | Havrix 720 | IC51, Subjects Aged >= 2 Months to <1 Year | Prevnar
Number analyzed (Participants) | 1280 | 394 | 131 | 64
percentage of participants
  Rate of subjects with SAE | 0.5 [0.2 to 1.0] | 1.0 [0.3 to 2.6] | 0 [0 to 2.8] | 1.6 [0 to 8.4]
  Rate of subjects with medically attended AE | 16.1 [14.1 to 18.2] | 14.2 [10.9 to 18.1] | 38.2 [29.8 to 47.1] | 42.2 [29.9 to 55.2]

5. Secondary Outcome: Rate of Subjects With Solicited Local and Systemic AEs
Description: Rate of subjects with solicited local and systemic AEs. Solicited AEs of local and systemic tolerability, i.e., reactions at the injection site or systemic reactions typical for vaccinations, were to be evaluated for 7 consecutive days after each vaccination (except after the HAVRIX®750 and Prevnar® injections at Month 7 [Visit 4]) and recorded in the subject diary.
  For this analysis IC51 vaccine recipients are displayed by age group rather than by dose group. This allows comparison of the safety profile of IC51 with the active control for the respective age group: Prevnar for study participants aged >= 2 months to <1 year and Havrix 720 for study participants aged >= 1 year.
Time Frame: 7 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Havrix 720: Havrix®720 0.5 ml im. at day 0 and month 7; Havrix®720 0.5 ml im. at day 0 and month 7; active comparator for subjects aged ≥1 to <18 years
Arm/Group | IC51, Subjects Aged >= 1 Year | Havrix 720 | IC51, Subjects Aged >= 2 Months to <1 Year | Prevnar
Number analyzed (Participants) | 1280 | 394 | 131 | 64
percentage of participants | 40.8 [38.1 to 43.5] | 29.4 [25.0 to 34.2] | 58 [49.1 to 66.6] | 59.4 [46.4 to 71.5]

6. Secondary Outcome: Rate of Subjects With Unsolicited AEs up to Day 56 and up to Month 7
Description: Rate of subjects with unsolicited AEs up to Day 56 and up to Month 7; For this analysis IC51 vaccine recipients are displayed by age group rather than by dose group. This allows comparison of the safety profile of IC51 with the active control for the respective age group: Prevnar for study participants aged >= 2 months to <1 year and Havrix 720 for study participants aged >= 1 year.
Time Frame: Day 56 and up to Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IC51, Subjects Aged >= 1 Year | Havrix 720 | IC51, Subjects Aged >= 2 Months to <1 Year | Prevnar
Number analyzed (Participants) | 1280 | 394 | 131 | 64
percentage of participants
  Day 56 | 46.5 [43.7 to 49.3] | 46.4 [41.4 to 51.5] | 72.5 [64.0 to 80.0] | 65.6 [52.7 to 77.1]
  Month 7 | 58.5 [55.8 to 61.2] | 57.6 [52.6 to 62.5] | 77.1 [68.9 to 84.0] | 81.3 [69.5 to 89.9]

7. Secondary Outcome: Rate of Subjects With Abnormal Laboratory Parameters
Description: Rate of subjects with abnormal laboratory parameters clinically significant results are shown below
Time Frame: Day 56 and Month 7
Population: Urinalysis Evaluations were not mandatory unless the subject was at least 12 years old at V0.
Measure: Number; unit: participants
Arm/Group | IC51 0.25 mL | IC51 0.5 mL | Havrix 720 | Prevnar
Number analyzed (Participants) | 871 | 540 | 394 | 64
participants
  Hemoglobin Day 56: number analyzed (Participants) | 831 | 536 | 391 | 47
  Hemoglobin Day 56 | 1 | 1 | 0 | 0
  Hemoglobin Month 7: number analyzed (Participants) | 821 | 531 | 386 | 47
  Hemoglobin Month 7 | 0 | 2 | 1 | 0
  Hematocrit Day 56: number analyzed (Participants) | 831 | 536 | 391 | 47
  Hematocrit Day 56 | 1 | 2 | 0 | 0
  Hematocrit Month 7: number analyzed (Participants) | 821 | 531 | 386 | 47
  Hematocrit Month 7 | 0 | 2 | 0 | 0
  White Blood Cells Day 56: number analyzed (Participants) | 831 | 536 | 391 | 47
  White Blood Cells Day 56 | 8 | 0 | 1 | 1
  White Blood Cells Month 7: number analyzed (Participants) | 821 | 531 | 386 | 47
  White Blood Cells Month 7 | 1 | 0 | 1 | 0
  Platelets Day 56: number analyzed (Participants) | 831 | 535 | 391 | 47
  Platelets Day 56 | 1 | 2 | 0 | 0
  Platelets Month 7: number analyzed (Participants) | 821 | 530 | 386 | 47
  Platelets Month 7 | 0 | 0 | 2 | 0
  Potassium Day 56: number analyzed (Participants) | 830 | 535 | 390 | 47
  Potassium Day 56 | 1 | 0 | 0 | 0
  Potassium Month 7: number analyzed (Participants) | 820 | 532 | 385 | 47
  Potassium Month 7 | 1 | 0 | 1 | 0
  Calcium Day 56: number analyzed (Participants) | 828 | 535 | 390 | 47
  Calcium Day 56 | 1 | 0 | 0 | 0
  Calcium Month 7: number analyzed (Participants) | 805 | 533 | 379 | 47
  Calcium Month 7 | 0 | 2 | 0 | 0
  AST Day 56: number analyzed (Participants) | 829 | 534 | 391 | 47
  AST Day 56 | 0 | 0 | 0 | 1
  AST Month 7: number analyzed (Participants) | 821 | 534 | 385 | 47
  AST Month 7 | 5 | 0 | 0 | 3
  ALT Day 56: number analyzed (Participants) | 830 | 534 | 391 | 47
  ALT Day 56 | 0 | 0 | 1 | 1
  ALT Month 7: number analyzed (Participants) | 821 | 534 | 385 | 47
  ALT Month 7 | 4 | 0 | 0 | 3
  Alkaline Phosphatase Day 56: number analyzed (Participants) | 829 | 535 | 391 | 47
  Alkaline Phosphatase Day 56 | 1 | 1 | 0 | 0
  Alkaline Phosphatase Month 7: number analyzed (Participants) | 821 | 534 | 385 | 47
  Alkaline Phosphatase Month 7 | 7 | 0 | 0 | 0
  Bilirubin Day 56: number analyzed (Participants) | 830 | 534 | 391 | 47
  Bilirubin Day 56 | 0 | 0 | 0 | 0
  Bilirubin Month 7: number analyzed (Participants) | 818 | 534 | 384 | 45
  Bilirubin Month 7 | 1 | 0 | 0 | 0
  Red Blood Cells Day 56: number analyzed (Participants) | 831 | 531 | 386 | 47
  Red Blood Cells Day 56 | 0 | 1 | 0 | 0
  Red Blood Cells Month 7: number analyzed (Participants) | 821 | 531 | 386 | 47
  Red Blood Cells Month 7 | 0 | 0 | 0 | 0
  Creatinine Day 56: number analyzed (Participants) | 827 | 533 | 390 | 47
  Creatinine Day 56 | 1 | 0 | 0 | 0
  Creatinine Month 7: number analyzed (Participants) | 818 | 532 | 385 | 47
  Creatinine Month 7 | 2 | 0 | 0 | 0
  Sodium Day 56: number analyzed (Participants) | 830 | 535 | 390 | 47
  Sodium Day 56 | 2 | 0 | 0 | 0
  Sodium Month 7: number analyzed (Participants) | 820 | 532 | 385 | 47
  Sodium Month 7 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months after first vaccination
Arm/Group | IC51 0.25 mL | IC51 0.5 mL | Havrix 720 | Prevnar
Serious Adverse Events (participants affected / at risk) | 16/871 | 7/540 | 10/394 | 1/64
Other Adverse Events (participants affected / at risk) | 691/871 | 300/540 | 252/394 | 57/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC51 0.25 mL (N=871) | IC51 0.5 mL (N=540) | Havrix 720 (N=394) | Prevnar (N=64)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 5 (5) | 0 (0) | 3 (3) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dengue Fever (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Typhoid Fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kawasaki´s Disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Familial Periodic Paralysis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IC51 0.25 mL (N=871) | IC51 0.5 mL (N=540) | Havrix 720 (N=394) | Prevnar (N=64)
Upper Respiratory Tract Infection (Infections and infestations) | 326 (414) | 67 (72) | 97 (115) | 33 (50)
Gastroenteritis (Infections and infestations) | 58 (61) | 3 (3) | 14 (14) | 9 (12)
Nasopharyngitis (Infections and infestations) | 77 (89) | 14 (16) | 27 (27) | 5 (6)
Pyrexia (General disorders) | 122 (127) | 35 (36) | 36 (40) | 8 (10)
Heat Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 4 (4) | 4 (4) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 30 (32) | 3 (3) | 10 (10) | 5 (5)
Rhinitis (Infections and infestations) | 45 (48) | 8 (8) | 17 (19) | 3 (5)
Injection Site Pain (General disorders) | 15/256 (17) | 65/532 (74) | 20/228 (20) | 0/0 (0) — pain without touching, solicited local
Tenderness (General disorders) | 38 (40) | 48 (55) | 27 (27) | 8/63 (10) — pain upon touching, solicited local
Hardening (General disorders) | 10 (10) | 8 (8) | 2 (2) | 5/63 (6) — solicited local
Swelling (General disorders) | 34 (35) | 14 (15) | 12 (15) | 5/63 (6) — solicited local
Redness (General disorders) | 81 (93) | 22 (22) | 25 (25) | 23/63 (30) — solicited local
Flu-like symptoms (General disorders) | 21/268 (23) | 16/532 (17) | 16/235 (16) | 0/0 (0) — solicited systemic
Headache (Nervous system disorders) | 10/233 (10) | 31/531 (37) | 10/219 (10) | 0/0 (0) — solicited systemic
Fever (General disorders) | 244 (316) | 61 (76) | 49 (53) | 24/63 (31) — solicited systemic
Irritability (General disorders) | 87 (111) | 6 (9) | 16 (17) | 9/63 (16) — solicited systemic
Vomiting (Gastrointestinal disorders) | 58 (69) | 10 (11) | 13 (14) | 5/63 (5) — solicited systemic
Diarrhea (Gastrointestinal disorders) | 94 (113) | 6 (6) | 13 (13) | 6/63 (7) — solicited systemic
Rash (Skin and subcutaneous tissue disorders) | 49 (57) | 5 (5) | 6 (6) | 9/63 (9) — solicited systemic
Loss of appetite (Metabolism and nutrition disorders) | 65 (78) | 11 (14) | 13 (16) | 6/63 (12) — solicited systemic
Excessive Fatigue (General disorders) | 28 (32) | 12 (14) | 5 (5) | 5/63 (7) — solicited systemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other